CLINICAL TRIAL: NCT04102748
Title: Evaluation of Esthetic Outcomes of M-flap Implant Uncovering Technique Versus I-shaped Incision Around Single Implants in the Anterior Maxilla Using Pink Esthetic Score (PES) (RCT)
Brief Title: Evaluation of Esthetic Outcomes of M-shaped Flap Implant Uncovering Technique Versus I-shaped Incision Around Single Implants in the Anterior Maxilla Using Pink Esthetic Score
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Ezzat Mousa, Principal Investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ezzat Implant Master Thesis
Record Dates: First submitted 2019-09-21; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Dental Implant Failed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional (Active Comparator)
  Interventions: Procedure: I-incision, M-flap and conventional implant exposure techniques
- I-incision (Active Comparator)
  Interventions: Procedure: I-incision, M-flap and conventional implant exposure techniques
- M-flap (Active Comparator)
  Interventions: Procedure: I-incision, M-flap and conventional implant exposure techniques

INTERVENTIONS:
Procedure: I-incision, M-flap and conventional implant exposure techniques — Implant uncovering in the second stage using 3 different exposure techniques

SUMMARY:
The aim of this study is to evaluate the soft-tissue profile around a single-tooth implant in the anterior maxilla utilizing the PES after implant uncovering using "M" flap versus I-shaped incision.The primary objective is evaluation of esthetic outcomes around implant using PES.

Hypothesis: The use of I-shaped incision exposure technique will result in better esthetic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osseointegrated dental implant in the anterior maxilla.
* Patients of 20 - 50 years
* Periodontally healthy patients.
* No intraoral soft and hard tissue pathology.
* No systemic condition that contraindicate surgical intervention.

Exclusion Criteria:

* Intraoral soft and hard tissue pathology.
* Heavy smokers more than 20 cigarettes per day.
* Patients with systemic disease that may affect normal healing.
* Psychiatric problems.
* Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
PES | 3 months
  Esthetic outcomes around implant

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided